CLINICAL TRIAL: NCT01445834
Title: Retrospective Study About the Age-stratified Outcome of Pelvic Floor Muscle Exercise for Stress (SUI), Mixed (MUI) and Urgency Urinary Incontinence (UUI) 2003-2008
Brief Title: Age-stratified Outcome of Pelvic Floor Muscle Exercise for Urinary Incontinence
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Principal Investigator, Cornelia Betschart, Attending Urogynecology, MD, University of Zurich
Other Study IDs: KEK-ZH2011/0299/0
Record Dates: First submitted 2011-09-23; First posted 2011-10-04 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Stress Urinary Incontinence; Urge Urinary Incontinence
Keywords: outcome of pelvic floor muscle physiotherapy; female; stress urinary incontinence; urgency urinary incontinence; mixed urinary incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress; Urinary Incontinence, Urge

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Incontinent women

SUMMARY:
In this retrospective study the outcome of pelvic floor muscle training in 150 women will be tested regarding patients reported satisfaction and achievement of the incontinence improvement.

Comparison of two age groups, controlled for BMI, parity and previous incontinence operations.

DETAILED DESCRIPTION:
Pelvic floor muscle exercise is an established conservative treatment for female urinary incontinence. Up to now, the investigators don't know whether treatment outcome in elderly women is as good as in younger premenopausal women. The International Incontinence Society states 2009: "There is no good evidence to date to suggest that "healthy" older women with urinary incontinence do not benefit from pelvic floor muscle training as much as younger women".

In this retrospective study the investigators analyze patient charts from 2003-2008 regarding subjective patients and physiotherapists reported outcome after physiotherapy as well as for objective parameters like the need of an incontinence surgery in the follow-up of at least 2 years.

Eligibility criteria are age younger than 50 years (premenopausal) and age older than 65 years and a urodynamically proven urinary incontinence. As incontinence forms the investigators include in this study the following three form: stress urinary incontinence, mixed urinary incontinence and urgency urinary incontinence.

ELIGIBILITY:
Inclusion Criteria:

* premenopausal women (<50 years) with urodynamically proven urinary incontinence
* postmenopausal women (>65 years) with urodynamically proven urinary incontinence
* 9 sessions of pelvic floor muscle exercise in a professional kinesiological setting inbetween 2003-2008
* follow up regarding need of incontinence operation up to June 2011

Exclusion Criteria:

* women aged 50-65 years with urodynamically proven urinary incontinence
* stool incontinence

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: women from a tertiary referral center with urodynamically proven incontinence willig to perform physiotherapy
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2011-06; Primary Completion 2011-10 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Patients reported outcome regarding their urinary incontinence | 2003-2009 (up to 6 years)

SECONDARY OUTCOMES:
Physiotherapists reported outcome after finishing the pelvic floor muscle training | 2003-2008 (up to 5 years)
need of incontinence surgery after conservative treatment in the follow up of at least 2 years | follow up of at least 2 years after physiotherapy that was performed between 2003-2008

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia Betschart, MD, Principal Investigator — University Hospital of Zürich